CLINICAL TRIAL: NCT05868707
Title: To Evaluate a Phase III Study of OH2 Versus Investigator-selected Salvage Chemotherapy or Best Supportive Care in Melanoma Patients Who Had Failed Standard Therapy
Brief Title: OH2 Injection in Melanoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-020
Record Dates: First submitted 2023-05-03; First posted 2023-05-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
Keywords: Oncolytic virus
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OH2 (Experimental): OH2: 10^7 CCID50/mL intratumoral injection, once every 2 weeks;
  Interventions: Drug: OH2
- Salvage chemotherapy or best supportive care (Active Comparator): Salvage chemotherapy (single or combined, including but not limited to dacarbazine, temozolomide, taxoid, or platinum) or best supportive care selected by the investigator
  Interventions: Drug: Salvage chemotherapy or best supportive care

INTERVENTIONS:
Drug: OH2 — Oncolytic Type 2 Herpes Simplex Virus
  Arms: OH2
Drug: Salvage chemotherapy or best supportive care — single or combined, including but not limited to dacarbazine, temozolomide, taxoid, or platinum
  Arms: Salvage chemotherapy or best supportive care

SUMMARY:
To evaluate the efficacy of OH2 injection in patients with unresectable or metastatic melanoma who have failed at least second-line standard therapy, using investigator-selected salvage chemotherapy or best supportive care (BSC) as controls.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old, male or female;
2. Stage III or stage IV melanoma that has been definitively diagnosed by pathology and/or cytology and has failed at least second-line standard therapy (including chemotherapy, immunotherapy, and targeted therapy for those with genetic mutations) (progression to unresectable or metastatic melanoma within 6 months after the end of adjuvant therapy or during adjuvant therapy, This adjuvant therapy can be considered as advanced first-line therapy) for patients with unresectable or metastatic melanoma;
3. The overall percentage of subjects with mucosal melanoma will not exceed 22%;
4. Eastern Oncology Consortium (ECOG) physical condition score ECOG 0 ~ 1;
5. The expected survival time is more than 3 months;
6. At least 4 weeks after completion of previous antitumor therapy (including chemotherapeutic/radiotherapy, targeted therapy, immunotherapy) (at least 2 weeks after completion of previous bone radiotherapy, at least 6 weeks after withdrawal of chemotherapy using nitrosourea and mitomycin), and have recovered from adverse reactions of previous treatment (≤ grade 1 or baseline, except hair loss), and 4 weeks after surgery for major surgery;
7. At least one measurable target lesion was present according to RECIST 1.1 criteria. There are lesions suitable for intratumoral injection. Measurable tumor lesions were defined as longest diameter ≥10 mm and scanning thickness less than 5.0 mm. For lymph node lesions, short diameter ≥15 mm.
8. Asymptomatic central nervous system metastases, or treated asymptomatic brain metastases, must be examined by computed tomography (CT) or magnetic resonance imaging (MRI) for no disease progression, stable for at least 3 months, and without steroid medication for at least 4 weeks;
9. No severe dysfunction of major organs; Laboratory tests meet the following criteria:

   1. WBC≥3.0×109 / L, ANC≥2.0×109 / L (no correction by granulocyte colony stimulating factor [G-CSF] or granulocyte macrophage colony stimulating factor [GM-CSF] within 14 days prior to screening), PLT≥100×109 /L (do not receive platelet infusion or thrombopoietin [TPO], thrombopoietin (TPO) receptor agonist or interleukin-11 [IL-11] within 14 days before screening), Hb≥90 g/L (do not receive blood transfusion or erythropoietin [EPO] correction within 14 days before screening);
   2. Blood BUN and blood creatinine within the range of 1.5 times the upper limit of normal value;
   3. TBIL≤ 1.5 times the upper limit of normal (total bilirubin <2×ULN in subjects with Gilbert syndrome, or total bilirubin <3×ULN in subjects with indirect bilirubin indicating extrahepatic cause of total bilirubin elevation);
   4. ALT and AST≤ 2.5 times the upper limit of normal value; Patients with liver metastases do not exceed 5 times the upper limit of normal;
   5. Normal coagulation function (PT, APPT within 1.5 times the upper limit of normal);
10. Female subjects of childbearing age must have tested serum-negative for pregnancy before receiving the first trial drug;
11. Female subjects of reproductive age and male subjects with partners of women of reproductive age received effective forms of contraception during and for 3 months after treatment;
12. For subjects with genital herpes, need 3 months after the end of herpes;
13. Voluntary signing of informed consent, expected compliance is good.

Exclusion Criteria:

1. Severe medical conditions, including uncontrolled diabetes with medication, severe infections requiring systematic treatment, and active digestive tract ulcers;
2. Clinically important cardiovascular and cerebrovascular diseases exist, including:

   * Severe or uncontrolled heart disease requiring treatment, congestive heart failure rated III or IV by the New York Cardiology Association, unstable angina that cannot be controlled by medication, myocardial infarction in the last 6 months, ECG QTc interval: Severe arrhythmias requiring medication (other than atrial fibrillation or paroxysmal supraventricular tachycardia) ≥450 milliseconds in men and 470 milliseconds in women;
   * Patients with heart stents in place within 6 months;
   * Inadequately controlled hypertension, systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg;
3. History of primary uveal melanoma or other malignancies within 5 years prior to treatment (except early resection of cervical carcinoma in situ and skin cancer in situ);
4. A large amount of pleural fluid or ascites with clinical symptoms or symptomatic management;
5. Bone metastases (stable metastases controlled by treatment can be ruled out) or the presence of active, clinical BMS;
6. Have an active autoimmune disease that has required systemic treatment within the past 2 years (e.g. with disease-regulating drugs, corticosteroids, or immunosuppressive drugs). Replacement therapy (such as thyroxine, insulin, or physiologic corticosteroid replacement for renal or pituitary insufficiency) does not count as systemic therapy;
7. A history of immunodeficiency (HIV antibody positive), or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
8. Patients with active hepatitis B or hepatitis C: HbsAg or HBCAB-positive patients with HBV DNA copy number positive (limit of quantitative detection is 500IU/ml); HBV DNA (negative for HBV-DNA/below the hospital standard for quantitative testing) must be tested in the screening of such patients; Patients who tested positive for HCV antibodies were enrolled in this study only if HCV RNA test results were negative;
9. There is an active TB infection or other infectious disease that requires systematic treatment;
10. The subject has a known history of psychotropic substance abuse, alcoholism, or drug use;
11. Other investigational agents or antiviral therapies have been or are being used within 4 weeks prior to treatment, except for hepatitis B patients on ongoing treatment who may be treated with Entecavir, Tenofovir dipifuroxide fumarate, or adefovir dipivoxil;
12. Use of investigational drug within 4 weeks prior to initial dosing;
13. Had received live attenuated vaccine within 4 weeks prior to initial administration;
14. Pregnant or lactating women;
15. The investigator believed that the patient was not eligible to participate in the study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death from any cause，assessed up to 3 years
  Overall survival is defined as the interval from first dose to death from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Tumor assessments were performed every 8 weeks in first year and every 12 weeks thereafter until confirmed PD, start of new anticancer treatment, death, withdrawal of informed consent, loss of follow-up, or the end of the study, assessed up to 3 years
  Determination of the ORR is calculated based on the proportion of patients achieving CR or PR using the RECIST v1.1 and iRECIST as assessed by investigators.
Disease control rate (DCR) | Tumor assessments were performed every 8 weeks in first year and every 12 weeks thereafter until confirmed PD, start of new anticancer treatment, death, withdrawal of informed consent, loss of follow-up, or the end of the study, assessed up to 3 years
  DCR is defined as the percentage of participants with a best overall response of CR, PR, or SD.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Progression-free survival is defined as the time from first dose to the earlier event of confirmed PD or death from any cause.
Durable Response Rate (DRR) | Tumor assessments were performed every 8 weeks in first year and every 12 weeks thereafter until confirmed PD, start of new anticancer treatment, death, withdrawal of informed consent, loss of follow-up, or the end of the study，assessed up to 3 years
  DRR is defined as the percentage of participants with a best overall response of CR or PR using the RECIST/iRECIST assessment with a duration of response of at least 6 months.
Duration of Response (DOR) | Tumor assessments were performed every 8 weeks in first year and every 12 weeks thereafter until confirmed PD, start of new anticancer treatment, death, withdrawal of informed consent, loss of follow-up, or the end of the study，assessed up to 3 years
  DOR is defined as the time from the first recording of remission (CR or PR) to the first recording of disease progression or death (whichever comes first)

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hosptial, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hainan Cancer Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University and Hebei Tumor Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital ＆ Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute ＆ Hospital, Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital, Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Cancer Hospital Of The University Of Chinese Academy Of Sciences Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wang X, Tian H, Chi Z, Si L, Sheng X, Hu H, Gu X, Li S, Li C, Lian B, Zhou L, Mao L, Tang B, Yan X, Wei X, Li J, Liu B, Guo J, Kong Y, Cui C. Oncolytic virus OH2 extends survival in patients with PD-1 pretreated melanoma: phase Ia/Ib trial results and biomarker insights. J Immunother Cancer. 2025 Feb 6;13(2):e010662. doi: 10.1136/jitc-2024-010662. PMID 39915002